CLINICAL TRIAL: NCT04182607
Title: Donor Outcomes Following Hand-Assisted and Robotic Living Donor Nephrectomy: a Retrospective Review
Status: Recruiting | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 063.HPB.2019.D
Record Dates: First submitted 2019-11-27; First posted 2019-12-02 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-09

CONDITIONS: Transplant; Kidney Diseases
Keywords: kidney; transplant; nephrectomy
MeSH Terms: conditions — Kidney Diseases | interventions — Kidney Transplantation; Nephrectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- hand-assisted kidney transplant: Kidney donors and recipients who underwent a hand-assisted kidney transplant
  Interventions: Procedure: kidney transplant
- robotic kidney transplant: Kidney donors and recipients who underwent a robotic kidney transplant
  Interventions: Procedure: kidney transplant

INTERVENTIONS:
Procedure: kidney transplant — Clinical data will be collected from electronic medical records (EMRs) on donors and recipients who underwent a minimally invasive kidney transplantation procedure
  Other Names: nephrectomy

SUMMARY:
1.1. Background: Renal transplantation is the treatment of choice for eligible patients with end-stage renal disease. It provides better outcomes in terms of life expectancy and quality of life than dialysis (Liu, Narins, Maley, Frank, & Lallas, 2012). Kidney transplants from living donors also have additional benefits in terms of graft function and survival compared to transplants from cadaver donors (Galvani et al., 2012). Living donor transplants provide an opportunity to have good quality grafts and to perform the procedure when the recipient is in an optimal clinical status (Creta et al., 2019).

Laparoscopic donor nephrectomy was first introduced in 1995 and is currently accepted as the gold standard for kidney procurement from living donors. The first worldwide robotic assisted laparoscopic donor nephrectomy was performed in 2000 by Horgan et al. (Horgan et al., 2007).

The main obstacle to living donation is the exposure of a healthy subject to the risks of a major surgical intervention. Therefore, efforts have been made to reduce complications and postoperative pain, achieve faster recovery, and minimize the surgical incisions.

Minimally invasive procedures like hand-assisted and robotic approaches greatly enhance living donation rates, and in 2001 the number of living donors exceeded the number of cadaver donors (Horgan et al., 2007).

1.2. Aim(s)/Objective(s): The objective of this study is to compare intra- and postoperative patient outcomes of kidney donors following hand-assisted and robotic kidney transplants at a single center.

1.3. Rationale for the study: More research is needed regarding the differences between minimally invasive approaches to kidney transplantation.

DETAILED DESCRIPTION:
This is a retrospective, single-center cohort study. Clinical data will be collected from electronic medical records (EMRs) on donors and recipients who underwent a minimally invasive kidney transplantation procedure. Data from all patients who had a hand-assisted or robotic minimally invasive kidney transplantation procedure at Methodist Dallas Medical Center (MDMC) between January 2006 and November 2019 will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Kidney donors and recipients who underwent a hand-assisted or robotic kidney transplant

Exclusion Criteria:

* Patients that do not meet the Study Inclusion Criteria laid out above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data from all patients who had a hand-assisted or robotic minimally invasive kidney transplantation procedure at Methodist Dallas Medical Center (MDMC) between January 2006 and November 2019 will be included in the study
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2019-11-06 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Patient demographics | between January 2006 and November 2019
  Patient demographics of donors and recipients will be compared between surgical techniques (i.e., hand-assisted vs. robotic).
Kidney Laterality | between January 2006 and November 2019
  A chart review of which kidney (left versus right) was donated
operating room (OR) time (minutes) | between January 2006 and November 2019
  operating room (OR) time (minutes) of donors and recipients will be compared between surgical techniques (i.e., hand-assisted vs. robotic).
warm ischemia time (minutes) | between January 2006 and November 2019
  warm ischemia time (minutes) of donors and recipients will be compared between surgical techniques (i.e., hand-assisted vs. robotic).
estimated blood loss (EBL) (milliliters (mL)) | between January 2006 and November 2019
  estimated blood loss (EBL) of donors and recipients will be compared between surgical techniques (i.e., hand-assisted vs. robotic).
complications (using Clavien-Dindo scale) | between January 2006 and November 2019
  complications (using Clavien-Dindo scale) of donors and recipients will be compared between surgical techniques (i.e., hand-assisted vs. robotic).
hospital length of stay (LOS) (days from admit to discharge) | between January 2006 and November 2019
  hospital length of stay (LOS) (days from admit to discharge) of donors and recipients will be compared between surgical techniques (i.e., hand-assisted vs. robotic).
30-day readmissions | between January 2006 and November 2019
  30-day readmissions of donors and recipients will be compared between surgical techniques (i.e., hand-assisted vs. robotic).
BMI (kilogram per square meter (kg/m^2)) | between January 2006 and November 2019
  BMI (kilogram per square meter (kg/m^2)) of donors and recipients will be compared between surgical techniques (i.e., hand-assisted vs. robotic).
hospital-based charges/costs | between January 2006 and November 2019
  hospital-based charges/costs of donors and recipients will be compared between surgical techniques (i.e., hand-assisted vs. robotic).
creatinine levels at discharge (milligrams per deciliter (mg/dL)) | between January 2006 and November 2019
  creatinine levels at discharge (milligrams per deciliter (mg/dL)) of donors and recipients will be compared between surgical techniques (i.e., hand-assisted vs. robotic).

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Mejia, MD, Principal Investigator — The Liver Institute at Methodist Dallas Medical Center
Locations (1):
- The Liver Institute at Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will be accessed by the principal investigator and delegated staff only for the duration of the trial.